CLINICAL TRIAL: NCT00547742
Title: Correlation of PET-CT Studies With Serum Protein Analysis
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Dr Andrew Quon, Stanford University School of Medicine
Other Study IDs: VAR0011; 96184; VAR0011
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Carcinomas (Including Squamous Cell and Adenocarcinoma)
MeSH Terms: conditions — Carcinoma; Adenocarcinoma | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood

INTERVENTIONS:
Procedure: PET/CT Scan
Procedure: phlebotomy

SUMMARY:
To correlate serum proteomics patterns with PET/CT findings to improve cancer diagnosis, staging, prognosis, and therapy monitoring.

ELIGIBILITY:
Inclusion Criteria:1. Patients must have a PET/CT study performed at the time of blood collection.

2. Patients must understand and voluntarily sign an Informed Consent form after the contents have been fully explained to them. Exclusion Criteria:1. Patients who are not eligible for a PET/CT study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having PET/CT scans
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2005-07; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Andrew Quon, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States